CLINICAL TRIAL: NCT01732744
Title: A Castor Bean Solution Reduces Complete Denture Biofilm
Brief Title: A Castor Bean Solution for Cleaning Dentures
Acronym: ACBSFCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ingrid Machado de Andrade, Phd, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: FORP_491
Record Dates: First submitted 2012-09-26; First posted 2012-11-26 (Estimated); Last update posted 2012-11-26 (Estimated); Status verified 2012-11

CONDITIONS: Prostheses-related Infections
Keywords: biofilm, castor bean, sodium hypochlorite, alkaline peroxide
MeSH Terms: interventions — Saline Solution; Sodium Hypochlorite; Polident

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Physiological solution (Placebo Comparator): 1)Negative Control: physiological solution, for 20 minutes
  All the volunteers used one of the four chemical methods (interventions) in a random sequence for a period of 07 days each. Between each period of use, there was a one week wash out period during which the patient performed his/her habitual cleaning procedure, in order to avoid a carry-over effect.
  Interventions: Other: Physiological solution
- Sodium hypochlorite (Active Comparator): 2)active Comparator 1: Sodium hypochlorite, for 20 minutes
  All the volunteers used one of the four chemical methods (interventions) in a random sequence for a period of 07 days each. Between each period of use, there was a one week wash out period during which the patient performed his/her habitual cleaning procedure, in order to avoid a carry-over effect.
  Interventions: Other: Sodium hypochlorite
- Peroxide alkaline (Active Comparator): 2)Active Comparator 2: Alkaline peroxide (Polident), for 5 minutes
  All the volunteers used one of the four chemical methods (interventions) in a random sequence for a period of 07 days each. Between each period of use, there was a one week wash out period during which the patient performed his/her habitual cleaning procedure, in order to avoid a carry-over effect.
  Interventions: Other: Alkaline Peroxide
- Castor bean solution (Experimental): 3)Experimental: castor bean solution, for 20 minutes
  All the volunteers used one of the four chemical methods (interventions) in a random sequence for a period of 07 days each. Between each period of use, there was a one week wash out period during which the patient performed his/her habitual cleaning procedure, in order to avoid a carry-over effect.
  Interventions: Other: Castor bean solution

INTERVENTIONS:
Other: Physiological solution — The volunteers were instructed to brush the internal surface of complete dentures for 2 minutes, 3 times a day, after meals (breakfast, lunch and dinner) and use the following chemical immersion methods, only once a day after dinner: A - Control (Co): Physiological solution, for 20 minutes. B) 1% Sodium Hypochlorite, for 20 minutes. C) Polident Alkaline Peroxide, for 3 minutes. D) 2,0% Castor bean solution Ricinus communis, for 20 minutes. In addition, the participants were instructed to immerse their dentures in water during the night period, before going to sleep.
  Other Names: Saline solution
  Arms: Physiological solution
Other: Sodium hypochlorite — The volunteers were instructed to brush the internal surface of complete dentures for 2 minutes, 3 times a day, after meals (breakfast, lunch and dinner) and use the following chemical immersion methods, only once a day after dinner: A - Control (Co): Physiological solution, for 20 minutes. B) 1% Sodium Hypochlorite, for 20 minutes. C) Polident Alkaline Peroxide, for 3 minutes. D) 2,0% Castor bean solution Ricinus communis, for 20 minutes. In addition, the participants were instructed to immerse their dentures in water during the night period, before going to sleep.
  Other Names: 1% Sodium hypochlorite
  Arms: Sodium hypochlorite
Other: Alkaline Peroxide — The volunteers were instructed to brush the internal surface of complete dentures for 2 minutes, 3 times a day, after meals (breakfast, lunch and dinner) and use the following chemical immersion methods, only once a day after dinner: A - Control (Co): Physiological solution, for 20 minutes. B) 1% Sodium Hypochlorite, for 20 minutes. C) Polident Alkaline Peroxide, for 3 minutes. D) 2,0% Castor bean solution Ricinus communis, for 20 minutes. In addition, the participants were instructed to immerse their dentures in water during the night period, before going to sleep.
  Other Names: Effervescent tabs; Polident
  Arms: Peroxide alkaline
Other: Castor bean solution — The volunteers were instructed to brush the internal surface of complete dentures for 2 minutes, 3 times a day, after meals (breakfast, lunch and dinner) and use the following chemical immersion methods, only once a day after dinner: A - Control (Co): Physiological solution, for 20 minutes. B) 1% Sodium Hypochlorite, for 20 minutes. C) Polident Alkaline Peroxide, for 3 minutes. D) 2,0% Castor bean solution Ricinus communis, for 20 minutes. In addition, the participants were instructed to immerse their dentures in water during the night period, before going to sleep.
  Other Names: Ricinus communis solution; Castor oil solution
  Arms: Castor bean solution

SUMMARY:
To evaluate the efficacy of a castor bean-based solution (Ricinus communis) for removal of complete denture biofilm, comparing it with two products available on the market (sodium hypochlorite and alkaline peroxide). Fifty complete maxillary denture-wearers were instructed to brush their dentures after meals and once a day, for a period of 07 days, immerse them in the following solutions: A - Control: Physiological solution(20 minutes). B - Polident alkaline peroxide(3 minutes). C - 1% sodium hypochlorite(20 minutes). D - castor bean-based solution(20 minutes). The participants immersed their dentures in each of the solutions, according to a randomized sequence. For biofilm quantification, before (Baseline) and after the use of each product, the internal surfaces of maxillary complete dentures were revealed (1% neutral red), photographed and the stained biofilm was quantified with the aid of software (Image Tool 3.0). After concluding measurements of the areas (total and biofilm), the percentage of surface covered by biofilm of the complete denture was calculated .

DETAILED DESCRIPTION:
The study sought to minimize the occurrence of bias, and whenever possible sought to "blind" the parties involved (researchers, volunteers and statisticians), since none of them had knowledge of the allocation of treatments. The present study also followed the criteria described in the CONSORT Declaration

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders, age-range 45 years and over, completely edentulous, in a good state of general health, wearers of maxillary complete dentures fabricated of heat polymerized acrylic resin and acrylic artificial teeth.

Exclusion Criteria:

* Dentures that had been used for less than 03 years, and broken, fractured or relined dentures.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Denture area covered with biofilm | 8 weeks
  The volunteers were instructed to brush their dentures ,3 times a day and use the following chemical immersion methods, only once a day after dinner: A)Physiological solution .B) 1% Sodium Hypochlorite .C) Polident Alkaline Peroxide .D) 2,0% Castor bean solution . All the volunteers used one of the four chemical methods in a random sequence for a period of 07 days each. Between each period of use, there was a one week wash out period during which the patient performed his/her habitual cleaning procedure.On the first day and after 07 days of using the interventions, the internal surfaces of dentures were revealed with 1% neutral red solution and photographed with a digital photographic camera. Biofilm was measured on the photographic images of the complete dentures, using the computerized quantitative method "ImageTool". After concluding measurements of the areas (total and biofilm), the percentage of surface covered by biofilm of the complete denture was calculated .

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid M Andrade, PhD, Principal Investigator — University of Sao Paulo